CLINICAL TRIAL: NCT01826721
Title: Impact of an E-learning Tool on Patient Satisfaction, Knowledge and Medication Adherence in Solid Organ Transplantation: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Harrison (Other)
Responsible Party: Sponsor-Investigator, Jennifer Harrison, Pharmacy Clinical Site Leader, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: REB10-0987-AE
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Solid Organ Transplantation
Keywords: Solid organ transplantation; Immunosuppression; Education; E-learning; Medication knowledge; Patient satisfaction; Medication adherence
MeSH Terms: conditions — Patient Satisfaction; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Patients in the Standard of Care arm receive the usual in-hospital post-transplant medication teaching class led by a transplant pharmacist.
- TMITT (Active Comparator): Patients in this arm receive the standard of care plus the TMITT educational intervention.
  Interventions: Other: Transplant Medication Information Teaching Tool

INTERVENTIONS:
Other: Transplant Medication Information Teaching Tool — Online e-learning tool for post-transplant medication education.
  Arms: TMITT

SUMMARY:
Solid organ transplant recipients (SOTR) must follow complex medication regimens and require a substantial amount of education for effective self-management. The current standard of care for post-transplant medication teaching is a Self Medication education program conducted in hospital by the pharmacist. The Transplant Medication Information Teaching Tool (TMITT) is a web-based e-learning tool for SOTR developed at the Toronto General Hospital. The ability to control the content, sequence, pace and timing of education in order to achieve personal learning objectives, as well as the opportunity for ongoing review and reinforcement of information, may be an attractive, convenient and effective teaching modality.

SOTR will be randomly assigned to receive the standard of care or the standard of care plus the TMITT intervention. Primary objectives are to compare patient satisfaction and medication knowledge between the two groups at baseline and 3 months using modified versions of previously published questionnaires. Medication adherence as measured by a multidimensional approach including both subjective and objective components, will also be compared at 3 months. Our hypothesis is that an education strategy that includes both the standard pharmacist teaching followed by a tailored online e-learning intervention post-discharge will lead to improved patient satisfaction, knowledge and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing solid organ transplantation at Toronto General Hospital during the study period

Exclusion Criteria:

* non-English speaking/reading
* no internet access at home
* planned discharge to a rehab facility without internet access
* not on a calcineurin inhibitor (CNI) or sirolimus
* attending the Self Medication class on the same day as hospital discharge
* cognitive impairment that precludes participation in Self Medication program (as per the assessment of the transplant pharmacist)
* incapable of providing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Medication Knowledge Score from baseline to 3 months | Baseline and 3 months
  Medication Knowledge Score consists of 2 parts - recall of medication regimen and multiple choice knowledge questionnaire.

SECONDARY OUTCOMES:
Patient Satisfaction | Baseline and 3 months
  Patient satisfaction with medication information received.
Medication Adherence | 3 months
  Adherence to the immunosuppressant medication regimen is evaluated using the Multidimensional Adherence Classification System. This consists of patient self-report and measurement of standard deviation of immunosuppressant blood levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Harrison, BScPhm, MSc, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Harrison JJ, Badr S, Hamandi B, Kim SJ. Randomized Controlled Trial of a Computer-Based Education Program in the Home for Solid Organ Transplant Recipients: Impact on Medication Knowledge, Satisfaction, and Adherence. Transplantation. 2017 Jun;101(6):1336-1343. doi: 10.1097/TP.0000000000001279. PMID 27367473
- See also: Related Info — http://www.tmitt.ca